CLINICAL TRIAL: NCT02656485
Title: A Double Blind, Placebo-Controlled, Single Center, Randomized, Sequential, Ascending 14-Day Multiple Dose Study in Subjects With Acne Vulgaris to Evaluate the Safety, Tolerability and Preliminary Efficacy of B244 Delivered as a Topical Spray
Brief Title: A Double Blind, Placebo-Controlled, Randomized Study in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVB244-001
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose I (Experimental): B244 Dose 1 (dose level [cells/mL] 20,000,000,000)
  Interventions: Drug: B244; Drug: Placebo
- Dose II (Experimental): B244 Dose 2 (dose level [cells/mL] 40,000,000,000)
  Interventions: Drug: B244; Drug: Placebo
- Dose III (Experimental): B244 Dose 3 (dose level [cells/mL] 80,000,000,000)
  Interventions: Drug: B244; Drug: Placebo
- Placebo (Placebo Comparator): Placebo to Match B244
  Interventions: Drug: B244

INTERVENTIONS:
Drug: B244 — 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
Drug: Placebo — 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
  Arms: Dose I; Dose II; Dose III

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled study in subjects with acne vulgaris.

DETAILED DESCRIPTION:
After a screening visit and a one-week washout (if applicable), three sequential ascending doses of the study drug will be applied twice-daily (BID) for 14 days in three groups of subjects. Each group of subjects will be randomized to receive the planned doses of B244 or placebo BID

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 and ≤45 years of age
2. In good general health as determined by a thorough medical history and physical examination, electrocardiogram (ECG), vital signs, and clinical laboratory evaluation. Results of clinical laboratory tests must be without clinically significant abnormalities, including hematology, clinical chemistry and urinalysis.
3. Clinical diagnosis of facial acne vulgaris defined as:

   * ≥105 inflammatory lesions
   * ≥10 non-inflammatory lesions
   * IGA ≥2
4. Willing to refrain from using any treatments, other than the investigational product, including antibiotics, for acne present on the face. Topical acne treatments that do not have significant or measurable systemic absorption (e.g., benzoyl peroxide, salicylic acid) are allowed for treatment of acne of the back, shoulders and chest only.
5. Ability to comprehend and comply with procedures
6. Agree to commit to participate in the current protocol
7. Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read)

Exclusion Criteria:

1. Female subjects who are pregnant or lactating or who are trying to conceive
2. Female subjects with a positive urine β-human chorionic gonadotropin (β-hCG) test at screening or positive β-hCG urine at pre-dose
3. Any clinically relevant abnormality identified on the screening history, physical or laboratory examinations, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
4. Any skin condition which may interfere with the evaluation of safety or of acne vulgaris (e.g., rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne or folliculitis)
5. Use of tanning booths or excessive sun exposure, in the opinion of the investigator
6. Active cystic acne or acne congoblata, acne fulminans, and secondary acne
7. Two or more active nodular lesions
8. Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to baseline
9. Treatment with systemic corticosteroids (including intranasal and inhaled corticosteroids) within 4 weeks prior to baseline
10. Treatment with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 4 weeks prior to baseline
11. Prescription topical retinoid use on the face within 4 weeks of baseline (e.g., tretinoin, tazarotene, adapalene)
12. Treatment with hormonal therapy or dose change to hormonal therapy within 12 weeks prior to baseline. Dose and frequency of use of any hormonal therapy started more than 12 weeks prior to baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, estrogenic and progestational agents such as birth control pills.
13. Use of androgen receptor blockers (such as spironolactone or flutamide)
14. Oral retinoid use (e.g., isotretinoin) within 12 months prior to baseline or vitamin A supplements greater than 10,000 units/day within 6 months of baseline
15. Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the 8 weeks of the first dose or during the study
16. A positive urine drug screen for drugs of abuse, including alcohol or positive urine cotinine (≥300 ng/mL for cotinine) at the screening visit or at entry to the clinic (Note: urine cotinine required at screening visit only)
17. Treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of the screening period (this includes investigational formulations of marketed products, inhaled and topical drugs)
18. Hypersensitivity to B244 or its components
19. Blood collection of greater than 500 mL within 56 days prior to screening
20. Seropositive for human immunodeficiency virus (HIV) at screening
21. Positive for Hepatitis B virus surface antigen (HBsAg) or positive Hepatitis C virus antibody (HCV Ab) at screening
22. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hino, MD, Principal Investigator — Stephens Associates
Locations (1):
- Stephens Associates, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose I: BB244 Dose I : 10 pumps of spray applied BID twice a day to the entire face for 14 days
- Dose II: BB244 Dose II : 10 pumps of spray applied BID twice a day to the entire face for 14 days
- Dose III: BB244 Dose III: 10 pumps of spray applied BID twice a day to the entire face for 14 days
- Placebo: Placebo: 10 pumps of spray applied BID twice a day to the entire face for 14 days
Period: Overall Study
Arm/Group | Dose I | Dose II | Dose III | Placebo
Started | 9 | 9 | 9 | 9
Completed | 7 | 6 | 7 | 7
Not Completed | 2 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All subjects were adult men or women, between the ages of 18 and 45 years.
Groups:
- Dose I: B244 dose strength I
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Dose II: B244 dose strength II
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Dose III: B244 dose strength III
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Placebo: Placebo
  Placebo: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Total: Total of all reporting groups
Arm/Group | Dose I | Dose II | Dose III | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.0) | 26 (8.2) | 29.2 (4.8) | 31.7 (10.1) | 29.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 7 | 9 | 28
  Male | 2 | 4 | 2 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 2 | 7
  White | 3 | 2 | 5 | 4 | 14
  More than one race | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 3 | 3 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety (Number of Participants With Treatment Related Adverse Events)
Description: Number of participants with treatment related adverse events as assessed by physical examination, vital signs, clinical laboratory values, local skin responses
Time Frame: 4 weeks
Population: The safety analysis set included all subjects in the ITT/Safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Dose I: B244 dose I
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Dose II: B244 dose II
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
- Dose III: B244 dose III
  B244: 10 pumps (1.4 ml) of spray must be applied BID twice a day to the entire face for 14 days
Arm/Group | Dose I | Dose II | Dose III | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 4 | 1 | 2 | 2

2. Secondary Outcome: Efficacy
Description: Absolute Change from Baseline in Total Number of Lesions
Time Frame: Baseline and 4 weeks
Population: All efficacy and safety data were analyzed using the ITT/Safety population.
Measure: Mean (Standard Deviation); unit: Lesions
Groups:
- Pooled Active Doses: Pooled Active Doses (Doses I, II, III)
- Placebo: Placebo Arm
Arm/Group | Pooled Active Doses | Placebo
Number analyzed (Participants) | 26 | 8
Lesions | -9.6 (12.09) | -6.7 (10.66)

ADVERSE EVENTS:
Time Frame: Subjects were monitored for Adverse Events from Study Day 1 through Day 28 of the study
Description: During each visit, the Investigator questioned the subject about adverse events using an open question taking care not to influence the subject's answers, e.g., "have you noticed any change in your health?"
Arm/Group | Dose I | Dose II | Dose III | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 1/9 | 2/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose I (N=9) | Dose II (N=9) | Dose III (N=9) | Placebo (N=9)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Application Site Pain (General disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary Tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Streptococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No